CLINICAL TRIAL: NCT05685576
Title: Evaluation of a Combined Ridge Expansion Technique With Simultaneous Dental Implant Placement in Narrow Posterior Mandible
Brief Title: Evaluation of a Combined Ridge Expansion Technique With Simultaneous Dental Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lydia Nabil (Other)
Responsible Party: Sponsor-Investigator, Lydia Nabil, Associate Professor of Oral and Maxillofacial Surgery, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAlexandriaDentSurg22
Record Dates: First submitted 2023-01-04; First posted 2023-01-17 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Alveolar Process Atrophy
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ridge splitting and osseodensification with simultaneous implant placement (Experimental)
  Interventions: Device: Piezotomed ridge splitting and osseodensification

INTERVENTIONS:
Device: Piezotomed ridge splitting and osseodensification — Ridge expansion using piezotomed ridge splitting and osseodensification

SUMMARY:
Patients with long span, narrow edentulous ridge in the posterior mandible underwent piezotomed ridge splitting and osseodensification with simultaneous implant placement.

DETAILED DESCRIPTION:
This study is a single arm clinical trial. Patients of both genders, who are indicated for ridge splitting, were recruited from the outpatient clinic, Faculty of dentistry, Alexandria University.

The PICO question: "What is the effect of piezotomed ridge splitting and osseodensification on implant placement in narrow posterior mandibular ridges?"

Ethical approval for the study was obtained from the regional Ethical Review Board of the Faculty of Dentistry. All patients were informed about the procedure details, and each participant signed a written consent.

Ridge expansion was accomplished by piezotomed ridge splitting and osseodensification. Simultaneous implant placement was done in the same procedure.

Implant stability was assessed. Also, bone width gained and bone density were measured around the dental implants using cone beam computed tomography.

ELIGIBILITY:
Inclusion Criteria:

* Patients with good oral hygiene
* Patients with long-span, narrow posterior edentulous mandibular area
* Age limit range [25 - 66 years]
* Patients who accept to participate in the study
* Minimum height 10mm from the crest of the ridge till the upper border of inferior alveolar canal
* Minimum ridge thickness = 3mm at the crestal region
* If the patient is diabetic, should be controlled.

Exclusion Criteria:

* Immunosuppressive/ autoimmune disease patients
* Patients with osteoporosis
* Lack of sufficient amount of keratinizing mucosa at the crest of the edentulous saddle
* Patients with bleeding disorder disease
* Ridge width less than 3 mm
* Smokers
* Patients having periodontal disease
* The presence of a pathological lesion in the area of ridge splitting

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2023-03-05 (Actual)

PRIMARY OUTCOMES:
The score of primary implant stability | immediately at time of implant insertion
  - Primary stability of the implants is measured using:
  * insertion torque and
  * resonance frequency analysis by Osstell ISQ device (Osstell ISQ, W&H, Sweden)

SECONDARY OUTCOMES:
The width of bone gained | 3 months postoperative
  Width of bone gained at the crest of the ridge is measured by cone beam computed tomography in mm
The mean bone density around dental implants | 3 months postoperative
  The mean bone density around dental implants is measured by cone beam computed tomography in grey scale values

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No